CLINICAL TRIAL: NCT03323775
Title: Sensory Mapping of Lumbar Facet Joint Pain
Acronym: SENS-MAP
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2/107/17
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Chronic Pain; Facet Joint Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Suprathreshold stimulation — Intraoperatively, radiofrequency needles will be placed on specific nerves targeted using parallel needle placement technique under image guidance. These nerves will have identified by the diagnostic injections carried out previously. The nerves will be located using 50 Hz sensory stimulation. The targeted medial branches (dorsal ramus in the case of L5) will be stimulated using suprathreshold stimulation (up to three times the sensory detection threshold) to identify the pain referral area. Motor stimulation of 2 Hz will be used to identify the multifidus muscle as well as to evaluate the close proximity to major spinal nerve to improve the safety of the procedure.

SUMMARY:
Low back pain is a major contributor to the chronic pain burden in the community. Although there are numerous pain generators in the spine, lumbar facet joints are one of the most common sources of pain. A variety of measures such as physiotherapy, oral analgesics and minimally invasive injections are used to treat lumbar facet joint pain.

Facet joint steroid injections and radiofrequency denervations of the facet joint are the most commonly performed minimally invasive pain procedures for lumbar facet joint pain. Radiofrequency denervation is carried out by thermal lesioning of the medial branches that supply the facet joints. Conventionally two medial branches have been shown to innervate one facet joint and based on this, the norm is to lesion two nerves to denervate one facet joint. However, there is some variation in the nerve supply which may account for failure or false negative results of the diagnostic blocks.

The aim of the present study is to explore the feasibility of sensory mapping, thereby referral pattern of the lumbar medial branches using suprathreshold stimulation and to correlate the referral patterns with painful areas in the back and leg. It will also test if the present method of lesioning two nerves to denervate one facet joint is appropriate.

DETAILED DESCRIPTION:
Chronic pain is defined as pain lasting more than three months duration. Between one third and one half of the population of the UK are affected by chronic pain. This corresponds to just less than 28 million adults. Chronic low back pain is an important contributor to the chronic pain burden. Up to a third of UK's population is affected by low back ache each year and 20% visit their general practitioner for advice. The result is that nearly 2.6 million people are seeking medical care for back pain in a year. This translates into a huge economic burden on the already stretched healthcare budgets. The health care cost of low back ache was estimated to be £1632 million in 1998.4 However the indirect cost of low back pain mainly due to lost productivity is much higher and conservative estimates put it at £3440 million in 1998. It would not be hard to imagine what the present economic burden of chronic low back pain would be if inflation is factored in to the above figures. Apart from the fact that chronic low back pain has a huge economic impact, it does cause significant loss of function from an individual's perspective, damaged relationships and difficulties at workplace.

Lumbar facet joint pain

Mechanical low back pain is the most common cause of chronic low back pain. Anatomical structures, such as facet joints, sacro-iliac joints, posterior longitudinal ligaments and muscles have been found to generate and contribute to the mechanical low back pain. The lumbar zygapophyseal (facet) joints are the pain generators in 15% to 45% of patients with chronic low back pain. Variety of interventional treatment modalities have been used to treat facet joint pain. Intraarticular injections of steroids and radiofrequency (RF) ablation of the nerve supply of the facet joints are the most widely practised. A recent NICE guideline (NG 59) has recommended radiofrequency denervation but not steroid injections for proven lumbar facet joint pain.

The lumbar facet joints are innervated by the medial branches of posterior primary ramus of the spinal nerve (L1-L5). Each of these posterior primary rami divide into medial, intermediate and lateral branches (except L5 posterior primary ramus). The medial branches innervate the facet joints and the multifidus muscle. The intermediate branches innervate the muscle longissimus thoracis. The lateral branches innervate the iliocostalis lumborum muscle. The lateral branches of L1, 2 ,3 supply the skin over the lower back.

The nerve supply - medial branch and dorsal ramus have been the target for RF interventions to relieve facet joint pain. Anatomical studies in 1980s found that facet joint has a dual innervation - for instance, the L4-5 facet joint derives its innervation from the medial branches of dorsal rami of L3 and L4. The medial branches of L1-4 and the posterior primary ramus of L5 have a relatively fixed anatomical course, thereby rendering themselves good targets for interventions. This forms the basis of targeting two nerves to denervate one facet joint. The success rate of RF denervation varies from 50 to 90% .9, 10 The varied success rate is often attributed to single diagnostic blocks and procedural variations. But anatomical variation is not often considered. A recent study has showed that there is significant variation in the individual nerve supply to facet joints which may add to the false -negatives of diagnostic blocks and inadequate pain relief from radiofrequency denervation. One way of improving the success rate is to reproduce the pain by electrical stimulation prior to RF treatment.

Lumbar medial branches and fifth lumbar dorsal ramus have been electrically stimulated not only in healthy volunteers but also in pain patients. A recent study has shown that supratheshold stimulation of facet joints in healthy volunteers results in local and referred pain.However none of the studies have correlated the suprathreshold stimulation to map the painful area. Hence we propose to map the painful area by suprathreshold stimulation.

Rationale for Study Based on conventional anatomical studies, two medial branches are denervated to treat pain from one facet joint. But this does not take into account of the anatomical variation of individuals, thereby potentially over or under treating the pain. In this study the investigators will map the painful areas by stimulating the medial branches, thus estimating how necessary it is to lesion the medial branches according to the standard practice.

ELIGIBILITY:
Inclusion Criteria:

-Patients scheduled for radiofrequency denervation of lumbar medial branches and L5 dorsal ramus after adequate response to diagnostic testing

Exclusion Criteria:

* Unable to understand and comprehend the information given in English
* Inability to complete pain diagram

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants will be identified from the patients scheduled to undergo lumbar medial branch RF denervation at the surgical short stay unit, Aberdeen Royal Infirmary.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Stimulation of the target nerves. | Up to one hour after stimulation
  Self reported estimate of percentage coverage of pain reproduction by stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Aberdeen/NHS Grampian, Aberdeen, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No